CLINICAL TRIAL: NCT03471559
Title: Cannabidiol as a Medication for Neuropsychiatric and Other Medical Conditions - an in Vivo Innovative Drug Delivery Study
Brief Title: Cannabidiol - an in Vivo Innovative Drug Delivery Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Two step study, step two was not feasible based on results from phase one.
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CBD-DDS
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Pharmacokinetics, Bioavailability
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference formulation (Active Comparator): Cannabidiol capsule, 200 mg
  Interventions: Drug: Cannabidiol
- New formulation (Experimental): Cannabidiol, intranasal gel (XX mg, dose need to be determined during the study)
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — single or multiple dosing

SUMMARY:
Basic characterization of the drug delivery system for cannabidiol. A comparative bioavailability study.

DETAILED DESCRIPTION:
This study aims to investigate an innovative pharmaceutical preparation of cannabidiol. Thus, a comparative bioavailability study will be conducted, comparing cannabidiol capsules (reference formulation) with an intranasal cannabidiol gel (test formulation), with the further aim to find an appropriate dosing of the new pharmaceutical preparation. The intranasal administration may also be suitable to reduce the high variability in the bioavailability of cannabidiol observed for the current oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given by the subject
* Negative drug screening at the time of screening
* Non-smoking
* In female participants in fertile age, reliable contraception, which means contraception's Pearl index is equal to or smaller than 1.
* Body Mass Index between 18.5 kg/m2 and 30 kg/m2

Exclusion Criteria:

* Lack of accountability
* Pregnancy or lactation phase in females at the time of screening
* Any known psychiatric or neurological illness in the participant's history.
* Known family history regarding psychiatric disorders with an increased lifetime risk for psychiatric disorders in the participant (investigators qualified judgement)
* Relevant use of cannabis (which is defined on the present state of knowledge as more than five times lifetime consumption and/or more than two consumptions during the last year)
* Consumption of any illicit drugs (except cannabis in history, see above)
* Severe physical (internal) or neurological illness, especially cardiovascular, renal, advanced respiratory, haematologic or endocrinologic disorders or infectious diseases (acute hepatitis A, B or C or HIV) assessed at the time of the screening by the subject's history, clinical examination and laboratory testing, as assessed by the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of single dose - area under the curve (AUC(0-t)), AUC(0-∞)) | 36 hours
  reference formulation compared to new formulation
Pharmacokinetic profile of single dose - residual area | 36 hours
  reference formulation compared to new formulation
Pharmacokinetic profile of single dose - maximum concentration (Cmax) | 36 hours
  reference formulation compared to new formulation
Pharmacokinetic profile of single dose - time to reach Cmax (tmax) | 36 hours
  reference formulation compared to new formulation
Pharmacokinetic profile of single dose - elimination half life (t1/2) | 36 hours
  reference formulation compared to new formulation
Pharmacokinetic profile of single dose - elimination rate constant (λz) | 36 hours
  reference formulation compared to new formulation
Pharmacokinetic profile of multiple dosing - area under the curve (AUC(τ)) | 9 days
  reference formulation compared to new formulation
Pharmacokinetic profile of multiple dosing - maximum concentration (Cmax,ss) | 9 days
  reference formulation compared to new formulation
Pharmacokinetic profile of multiple dosing - time to reach Cmax (tmax,ss) | 9 days
  reference formulation compared to new formulation
Pharmacokinetic profile of multiple dosing - elimination half life (t1/2,ss (τ=12h)) | 9 days
  reference formulation compared to new formulation
Pharmacokinetic profile of multiple dosing - steady state accumulation ratio | 9 days
  reference formulation compared to new formulation

SECONDARY OUTCOMES:
Regular laboratory testing | 36h or 9 days
  standard laboratory blood tests
Electrocardiography - QTc time | 36 hours or 9 days
Vital signs - body temperature | 36 hours or 9 days
Vital signs - blood pressure | 36 hours or 9 days
  Systolic and diastolic blood pressure reported in millimetres of mercury (mmHg)
Vital signs - pulse rate | 36 hours or 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Fuhr, MD, Principal Investigator — Department I of Pharmacology, University of Cologne
Locations (1):
- Department I of Pharmacology, University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No